CLINICAL TRIAL: NCT06655506
Title: Enhanced Recovery Protocols in Gynecological Cancer Patients: a Feasibility Study
Brief Title: Enhanced Recovery Protocols in Gynecologic Oncology
Acronym: ERGO
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: University of Thessaly (Other); Aristotle University Of Thessaloniki (Other); Metaxa Hospital (Other); Saint Savvas Anticancer Hospital (Other)
Responsible Party: Principal Investigator, Nikolaos Thomakos, MD, PhD, MSc, Associate Professor of Obstetrics and Gynecology, National and Kapodistrian University of Athens
Other Study IDs: 131/2024
Record Dates: First submitted 2024-03-27; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: ERAS; Gynecologic Cancer; Perioperative Complication; Postoperative Pain; Quality of Life; Infections
MeSH Terms: conditions — Pain, Postoperative; Infections | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fulfilled ERAS criteria group: This group will include patients that achieved a compliance rate that exceeded 80% of the required predetermined criteria of ERAS protocols.
  Interventions: Combination Product: ERAS group
- Control group: This group will include patients that achieved a compliance rate that did not reach at least 80% of the required predetermined criteria of ERAS protocols.
  Interventions: Combination Product: Control group

INTERVENTIONS:
Combination Product: ERAS group — This group will include patients that achieved a compliance rate that exceeded 80% of the required predetermined criteria of ERAS protocols.
  Groups: Fulfilled ERAS criteria group
Combination Product: Control group — This group will include patients that do not follow the predetermined criteria of ERAS protocols
  Groups: Control group

SUMMARY:
Enhanced Recovery After Surgery (ERAS) are developed to provide a systematic structure for managing postsurgical patients.These protocols promote evidenced-based practices and implement a multidisciplinary effort to maintain normal physiology in the perioperative period and aid in earlier recovery. The present study aims to investigate the feasibility of and compliance to a structured ERAS protocol among Gynecological Oncological Centers in Greece as well as to compare the outcomes among patients that fullfilled the minimum number of necessary criteria, compared to those that were enrolled in ERAS protocols but did not meet the sufficient necessary criteria.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) are developed to provide a systematic structure for managing postsurgical patients.These protocols promote evidenced-based practices and implement a multidisciplinary effort to maintain normal physiology in the perioperative period and aid in earlier recovery. ERAS protocols briefly include pre-admission education, pre-operative nutritional care, specific recommendations for pre-operative medications, a standardized anesthetic protocol, perioperative fluid management, multimodal analgesia (MMA), early mobilization, and early removal of urinary catheters.

ERGO study study aims to investigate the feasibility of and compliance to a structured ERAS protocol among Gynecological Oncological Centers in Greece as well as to compare the outcomes among patients that fullfilled the minimum number of necessary criteria, compared to those that were enrolled in ERAS protocols but did not meet the sufficient necessary criteria. Patients will be registered into the trial before surgery. Quality assurance program will be in place for both patients that will fulfill the ERAS criteria as well as for those that will not fulfill them.

ELIGIBILITY:
Inclusion Criteria:

patients with gynaecological cancer and an ECOG performance status <4, ASA score <4.

Exclusion Criteria:

patients with metastatic cancer of non-gynaecological origin patients that are not able to follow ERAS protocol due to medical reasons patients with severe debilitating comorbidities (ECOG status 4, ASA score 4-5)

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is not based on self-representation
Study Population: In this study, patients that will be operated for gynecological cancer in the collaborating centers described in the Contacts and Locations section will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Duration of hospitalization | Up to 30 days postoperatively
  From date of hospitalization until the date of discharge or date of death from any cause, whichever came first, assessed up to 2 months.
Perioperative infections | Postoperatively (30 days)
  Number of participants with postoperative infections (including surgical site, pulmonary and urinary tract infections)

SECONDARY OUTCOMES:
Postoperative quality of life | Postoperatively (30 days)
  Documentation of quality of life using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C40) and the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaires. The EORTC-QLQ C30 involves 30 questions that are rated from 1 (no impact on quality of life) to 4 (debilitating symptoms). The FACT-G assesses physical, family, emotional and functional wellbeing through 27 questions that are scaled from 0 (no impact) to 4 (very much).
Postoperative morbidity (other than infectious) using the Clavien-Dindo classification | 30 days
  Major events such as pulmonary embolism,accuse myocardial infarction,etc
Interval to adjuvant therapy | Up to 100 days
  The interval between surgical treatment and adjuvant therapy (radiation and/or chemotherapytreatment) will be documented
Recurrence rates | 3 years follow-up
  Recurrent disease will be monitored through 3 year of follow up
Overall survival | 3 years follow-up
  Overall survival of the patients will be measured through 3 year of follow up

CONTACTS AND LOCATIONS:
Locations (8):
- Greece (8):
  - First department of Obstetrics and Gynecology, Athens, Athens
  - Agios Savvas Anticancer Hospital, Athens, Attica
  - First department of Obstetrics and Gynecology, National and Kapodistrian University of Athens, Athens, Attica
  - University of Thessaly, Larissa, Larissa
  - Metaxa Anticancer Hospital, Athens, Piraeus
  - Aristotle University of Thessaloniki, Second department of Obstetrics and Gynecology, Thessaloniki, Thessaloniki
  - Aristotle University of Thessaloniki, Third department of Obstetrics and Gynecology, Thessaloniki, Thessaloniki
  - Aristotle University of Thesalloniki, Papageorgiou Hospiral, Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
IPD will be provided upon reasonable request following communication with researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following study completion and up to 5 years from publication of findings.
Access Criteria: Data will be provided through a dedicated de-identified redcap database

REFERENCES:
- [Background] Pandraklakis A, Haidopoulos D, Lappas T, Stamatakis E, Valsamidis D, Oikonomou MD, Loutradis D, Rodolakis A, Bisch SP, Nelson G, Thomakos N. Thoracic epidural analgesia as part of an enhanced recovery program in gynecologic oncology: a prospective cohort study. Int J Gynecol Cancer. 2023 Nov 6;33(11):1794-1799. doi: 10.1136/ijgc-2023-004621. PMID 37652530
- [Background] Bogani G, Sarpietro G, Ferrandina G, Gallotta V, DI Donato V, Ditto A, Pinelli C, Casarin J, Ghezzi F, Scambia G, Raspagliesi F. Enhanced recovery after surgery (ERAS) in gynecology oncology. Eur J Surg Oncol. 2021 May;47(5):952-959. doi: 10.1016/j.ejso.2020.10.030. Epub 2020 Oct 28. PMID 33139130
- [Background] Nelson G. Enhanced Recovery in Gynecologic Oncology Surgery-State of the Science. Curr Oncol Rep. 2023 Oct;25(10):1097-1104. doi: 10.1007/s11912-023-01442-0. Epub 2023 Jul 25. PMID 37490193
- [Background] Nelson G, Fotopoulou C, Taylor J, Glaser G, Bakkum-Gamez J, Meyer LA, Stone R, Mena G, Elias KM, Altman AD, Bisch SP, Ramirez PT, Dowdy SC. Enhanced recovery after surgery (ERAS(R)) society guidelines for gynecologic oncology: Addressing implementation challenges - 2023 update. Gynecol Oncol. 2023 Jun;173:58-67. doi: 10.1016/j.ygyno.2023.04.009. Epub 2023 Apr 21. PMID 37086524
- [Background] Bhandoria GP, Bhandarkar P, Ahuja V, Maheshwari A, Sekhon RK, Gultekin M, Ayhan A, Demirkiran F, Kahramanoglu I, Wan YL, Knapp P, Dobroch J, Zmaczynski A, Jach R, Nelson G. Enhanced Recovery After Surgery (ERAS) in gynecologic oncology: an international survey of peri-operative practice. Int J Gynecol Cancer. 2020 Oct;30(10):1471-1478. doi: 10.1136/ijgc-2020-001683. Epub 2020 Aug 4. PMID 32753562
- [Derived] Pergialiotis V, Haidopoulos D, Daponte A, Tsolakidis D, Petousis S, Kalogiannidis I, Vlachos DE, Lygizos V, Fanaki M, Delinasios G, Tzitzis P, Ntailianas P, Theodoulidis V, Margioula Siarkou G, Daponte N, Thomakos N. Implementation Rates and Predictors of Compliance with Enhanced Recovery After Surgery Protocols in Gynecologic Oncology: A Prospective Multi-Institutional Cohort Study. Cancers (Basel). 2025 Dec 15;17(24):3991. doi: 10.3390/cancers17243991. PMID 41463241